CLINICAL TRIAL: NCT04048148
Title: A Double-masked, Randomized, Cross-over Comparative Study of Novel Myopia Control Designed Lens (Test Lens) Versus Single Vision Lens (SVL; Control)
Brief Title: Myopia Progression Trial With Novel Myopia Control Design Spectacle Lenses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brien Holden Vision Institute (Other)
Collaborators: Essilor International (Industry); Hai Yen Eye Care (Industry)
Responsible Party: Principal Investigator, Rebecca Weng, Senior Project Manager, Brien Holden Vision Institute
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: VCRTC2019-01
Record Dates: First submitted 2019-08-04; First posted 2019-08-07 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: This is a mono-center, randomized, double-masked, cross-over study to evaluate if novel design lens can slow down the progression of myopia. A total of 120 healthy children aged between 8 years to 13 years with myopia (-0.75D to -4.75D) meeting the inclusion and exclusion criteria will be recruited. These children will be randomized to wear test lenses followed by control lenses (Group 1) or to wear control lenses followed by test lenses (Group 2). At the end of the 12 month period, all participants will wear test lenses for another 6 months. All children will be followed at 3-monthly intervals for 1.5 years to monitor for changes in axial length and 6-monthly for changes in cycloplegic autorefraction. The cross-over design allows to compare treatment effects between the two groups at 6 months, 12 months and at 18 months. In addition, at the end of the study, the treatment effects can be compared within subject as each subject will have worn both lenses and serves as his/her control.
Who Masked: Participant, Investigator
Masking Description: Participants and their parents / guardians and investigators will be masked to their lens assignment. Test spectacles will be of similar appearance to control spectacles and will not be easily identified without specialized equipment. Test and control spectacles will be assigned a code (A or B) by the clinical coordinator and stored in a secure location.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novel myopia control lenses (Other): This group will be randomized to wear test lenses for 6 months followed by control lenses for 6 months and then test lenses for another 6 months
  Interventions: Device: Novel designed myopia control spectacle lenses
- Single vision lenses (Other): This group will be randomized to wear control lenses for 6 months followed by test lenses for 12 months
  Interventions: Device: Novel designed myopia control spectacle lenses

INTERVENTIONS:
Device: Novel designed myopia control spectacle lenses — A novel designed myopia control spectacle lenses (test lenses) will be given to both arms to wear for 12 months.

SUMMARY:
This is a mono-center, randomized, double-masked, cross-over study to evaluate rate of myopia progression with novel designed myopia control lens (test) compared to SVL (control). A total of 120 children will be recruited where 60 participants each will be randomized either to wear test (Group 1) or SVL lenses (Group 2) for 6 months each. At the end of the 6 months period, there will be a cross- over of lenses and the lenses evaluated for a further 6 months. At the end of the 12 month period, all participants (Group 1 and Group 2) will wear test lenses for another 6 months.

DETAILED DESCRIPTION:
Myopia has been considered as a 'global epidemic' owing to its rapid rise in prevalence across the world. Myopia significantly affects the quality of life of an individual socially by restriction of employment in various fields and economically by additional cost for eye care and spectacles and contact lenses (Lim, Gazzard et al. 2009). In addition, high myopia increases the risk of ocular morbidity such as retinal detachment, cataract, glaucoma which can could lead to blindness. Several optical and pharmaceutical strategies were developed over the recent years that could control or slow the progression of myopia.

It has been shown that persistent myopic defocus constantly applied on the whole retina has a beneficial effect on myopia progression, i.e. decrease in myopia progression (Anstice and Phillips 2011, Cheng, Woo et al. 2011, Ehsaei, Chisholm et al. 2011). In addition, a meta-analysis on the efficacy of non-invasive optical treatment strategies for myopia control reported prismatic bifocals to have the best outcome (Cheng, Woo et al. 2011). Therefore, test lenses were designed to increase the area and amount of myopic defocus on the retina without compromising vision.

Thus, this study aims to evaluate the efficacy of test lenses to reduce the progression of myopia by either reducing the myopia progression rate per year and/or reducing the elongation of eyeball through myopic defocus compared with SVL. A total of 120 healthy children aged 8 to 13 years will be recruited to participate in a double-masked cross-over clinical trial. Cycloplegic autorefraction will be the primary measure for myopia progression and axial length will the secondary outcome measure. Visual acuity will also be compared between test lens and control lens to determine the quality of vision using test lens.

ELIGIBILITY:
Inclusion Criteria:

General inclusion criterion:

- Volunteer subject and guardian, fluent Vietnamese spoken, willing to follow the protocol and able to read, comprehend and sign the informed consent form.

Study related inclusion criteria:

* Age: equal to or greater than 8 years and not older than 13 years.
* Spherical refractive error of -0.75 to -4.75 D in each eye (spherical equivalent), as measured by cycloplegic autorefraction.
* Astigmatism of not more than 1.50 D.
* Anisometropia of not more than 1.00 D.
* Best corrected visual acuity of equal or better than 0.05 LogMAR
* No strabismus by cover test at near and distance.
* Have the ability to comply with the protocol to get the reliable study measurements.
* Absence of ocular disease with full ophthalmic examination, such as retinal disease, cataract and ptosis. Good general health, without systemic or neurodevelopmental conditions. Without ocular or systemic medicine, which might affect myopia progression or visual acuity through known effects on retina, accommodation or significant elevation of intraocular pressure.
* No history of progressive addition lenses (PALs) or bifocal use and no prior use of contact lenses

Exclusion Criteria:

General exclusion criteria:

* Vulnerability of the subject,
* Participation in another study which might have an influence on vision or interfere with study assessments.

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 132 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Cycloplegic refraction | Up to 18 months
  Change in myopia progression measured by cycloplegic refraction (Diopters) using Shin Nippon Auto-refractor

SECONDARY OUTCOMES:
Axial length | Up to 18 months
  Change in ocular axial length (mm) measured using Lenstar Optical Biometer

CONTACTS AND LOCATIONS:
Overall Officials: Padmaja Sankaridurg, PhD, Study Director — Brien Holden Vision Institute
Locations (1):
- Hai Yen Eye Care, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Clinical study report will be shared once the study is completed. Study anticipate to be completed in 2020.
Supporting Information: CSR
Time Frame: The data will become available mid 2021, starting 6 months after publication.

REFERENCES:
- [Derived] Sankaridurg P, Weng R, Tran H, Spiegel DP, Drobe B, Ha T, Tran YH, Naduvilath T. Spectacle Lenses With Highly Aspherical Lenslets for Slowing Myopia: A Randomized, Double-Blind, Cross-Over Clinical Trial: Parts of these data were presented as a poster at the Annual Research in Vision and Ophthalmology meeting, 2022. Am J Ophthalmol. 2023 Mar;247:18-24. doi: 10.1016/j.ajo.2022.10.021. Epub 2022 Nov 5. PMID 36347276